CLINICAL TRIAL: NCT05696145
Title: Aortic Stenosis Associated Left Ventricular Remodeling - Impact of Genetic, Valvular and Non-valvular Factors
Brief Title: Aortic Stenosis Associated Left Ventricular Remodeling - An Investigation of Genetic and Gender Specific Differences in 170 Patients Undergoing Aortic Valve Replacement Surgery
Acronym: SALVAGE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Lisa Gundestrup (Other)
Responsible Party: Sponsor-Investigator, Lisa Gundestrup, MD., Odense University Hospital
Organization: Odense University Hospital (Other)
Other Study IDs: SALVAGE protocol version 1
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Aortic Valve Stenosis
Keywords: low flow low gradient aortic valve stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples + myocardial biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to investigate the genetic and gender specific differences, in patients with low flow low gradient aortic stenosis and high flow high gradient aortic stenosis. Patients referred for surgical aorticvalve replacement will be offered to participarte in the study.

The main questions the study aims to answer are:

1. Low-gradient aortic stenosis is associated with differences in valvular concentration of the genes that code for mast-cell chymase, Angiotensin-II, ACE, ACE2 and Angiotensin receptor 1 and 2.
2. Low-gradient aortic stenosis is associated with differences in the genetic code of renin-angiotensin-aldosterone system.
3. Gender differences in LV remodelling associates with different levels of sexual hormones.

Patients participating in the study will be asked to undergo:

* Cardiac ultrasound, MR- and CT-scan prior to surgery
* Blooddraw prior to surgery.
* Heartmuscle biopsy during surgery
* Cardiac MR-scan 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Severe AS (estimated by the local heart team, aortic valve area<1cm2) referred for AVR at the cardiology department at Odense University Hospital
2. Age > 18 years
3. Signed informed consent

Exclusion Criteria:

1. Bicuspid aortic valve.
2. LV systolic dysfunction (LVEF<50%).
3. Patients with concomitant moderate-severe aortic valve regurgitation.
4. Concomitant moderate-severe mitral valve regurgitation.
5. Moderate to severe nephropathy (s-creatinine >200 mmol/l)
6. Unwilling to participate in the study.
7. Claustrophobia.
8. Permanent cardiac devices (pacemaker and ICD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for surgical aortic valve replacement at the department of Cardiothoracic and vascular surgery at Odense University Hospital, Denmark will be evaluated and if they meet the inclusion criteria they will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Genetic polymorphisms betweem low flow low gradient and high flow high gradient aortic stenosis patients | At the time of surgery

IPD SHARING:
Plan to Share IPD: No